CLINICAL TRIAL: NCT02118610
Title: Treatment of Schizophrenia With L-tetrahydropalmatine (l-THP): a Novel Dopamine Antagonist With Anti-inflammatory and Antiprotozoal Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Deanna Kelly, Deanna L. Kelly, Pharm.D., BCPP, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HP-00058491
Record Dates: First submitted 2014-04-14; First posted 2014-04-21 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2022-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- l-tetrahydropalmatine (Experimental): l-tetrahydropalmatine (30 mg BID)
  Interventions: Drug: L-tetrahydropalmatine (30mg)
- Sugar Pill (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: L-tetrahydropalmatine (30mg) — Active comparator
  Arms: l-tetrahydropalmatine
Drug: Sugar pill — Placebo
  Arms: Sugar Pill

SUMMARY:
Schizophrenia is a devastating and complex illness, with multiple symptom and behavioral manifestations. Antipsychotic medications are the mainstay of treatment; however, many patients only partially respond to treatment. Development of new treatment has not progressed rapidly, in part, because the underlying etiopathophysiology of the illness is not well understood. To date, all pharmacological treatments approved for use in schizophrenia involve primary modulation of the dopamine system. Many agents without dopamine action have failed to demonstrate efficacy. There is growing evidence that schizophrenia may be, in part, due to an inflammatory process and pharmacological treatment approaches that decrease inflammation have shown promise. Thus, treatments that may have anti-inflammatory properties (e.g., TNF-alpha inhibition), but also possess dopamine modulation may prove to be beneficial. This novel medication, l-tetrahydropalmatine (l-THP), has robust anti-inflammatory properties, particularly TNF-alpha and ICAM inhibition; has antiprotozoal activity; and possesses an antipsychotic-like pharmacological profile of D1, D2 and D3 receptor antagonism. The high affinity of l-THP for D1 versus D2 receptors distinguishes it from first generation antipsychotics and its D1 to D2 ratio resembles that of the superior antipsychotic, clozapine. Also, an almost identical compound, l-stepholindine (l-SPD), demonstrates robust antipsychotic activity in humans (both positive and negative symptoms) and is currently used clinically in China. l-THP has been used for over 40 years clinically in China, has a good safety profile to date, and represents a novel and exciting mechanism for schizophrenia treatment. Initial safety data from our phase I study of l-THP (20 healthy controls) shows excellent tolerability and lack of any substantial side effects. L-THP has been tested in outpatient drug abuse trials for 4 weeks with good safety data, (Hu et al 2006, Yang et al 2003). Yang et al (2003) randomized this medication in over 120 participants for 4 weeks with 4 week observation without any notable side effects.

We will test this compound (30 mg BID) as an adjunct treatment in a randomized, double-blind, 4-week trial, in which we will assess treatment efficacy, changes in peripheral cytokine concentrations, and, secondarily, antiprotozoal effects, (antibody titers to Toxoplasma gondii), an infection that is known to occur at higher rates in schizophrenia than healthy controls and may be related in part to the illness.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-IV diagnosis of schizophrenia or schizoaffective disorder
2. Minimum score of 45 on the total Brief Psychiatric Rating scale or a CGI of 4
3. Age 18-64 years
4. Currently taking antipsychotic regimen with no dose changes in last 30 days
5. Ability to consent determined by a score of 10 or greater on the Evaluation to Sign Consent

Exclusion Criteria:

1. Women who are pregnant, nursing, or not using effective contraception (if capable of getting pregnant)
2. Current organic brain disorder or mental retardation
3. Medical condition whose pathology or treatment could alter the presentation or treatment of schizophrenia or significantly increase the risk associated with study medication. This includes HIV, kidney disease, congestive heart failure, pheochromocytoma, untreated hyperthyroidism, dehydration, fever, uncorrected congenital heart defect, seizures, electrolyte imbalance, uncontrolled diabetes mellitus, porphyria variegate, superventricular tachycardia, atrial fibrillation, cardiomyopathy, or cancer. This also may include other medical conditions where the medically accountable investigator in the study does not think it would be in the best interest of the participant to participate in the study.
4. Current (past month) substance abuse or dependence (DSM-IV criteria) other than nicotine or caffeine; substance use, per se, will not be exclusionary
5. Inability to provide valid informed consent
6. Inability to understand English
7. Inability to cooperate with study procedures
8. Taking herbal or homeopathic medications where the metabolism of the drug is not known

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2014-09; Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deanna L Kelly, Parm.D., BCPP, Principal Investigator — University of Maryalnd, Baltimore
Locations (1):
- Maryland Psyciatric Research Center, Catonsville, Maryland, United States

REFERENCES:
- See also: Maryland Psychiatric Research Center — http://www.mprc.umaryland.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | L-tetrahydropalmatine | Sugar Pill
Started | 30 | 33
Completed | 29 | 32
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L-tetrahydropalmatine | Sugar Pill | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 32 | 61
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (11.1) | 41.7 (10.1) | 41.65 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 20 | 23 | 43
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 18 | 17 | 35
  White | 9 | 13 | 22
  Other | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Symptom Improvement
Description: Measured by the Brief Psychiatric Rating Scale, positive symptom subfactor, Scale for the Assessment of Negative Symptoms (SANS) and Brief Negative Symptom Scale (BNSS).
  The total BPRS score is calculated by adding the scores for scales #1-#18. Each scale ranges from "1=Not Present" to "7=Very Severe". Total scores range from a minimum score of 18 to a maximum score of 126. A higher total score indicates a more severe psychiatric symptom rating.
Time Frame: Baseline and 4 weeks (endpoint)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-tetrahydropalmatine | Sugar Pill
Number analyzed (Participants) | 29 | 32
score on a scale
  Baseline | 41.3 (8.8) | 40.3 (6.9)
  Endpoint | 36.6 (9.0) | 37.3 (8.7)

2. Secondary Outcome: Improvement in Cognitive Function
Description: Neuropsychological testing will be done at baseline and endpoint using the MATRICS battery. A composite score as well as individual scores will be will be the outcome. This assessment total minimum score of -10 and maximum score of 80. The higher the score the better the outcome.
Time Frame: Baseline and 4 weeks (endpoint)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | L-tetrahydropalmatine | Sugar Pill
Number analyzed (Participants) | 29 | 32
score on a scale
  Baseline | 28.0 (13.9) | 27.7 (14.1)
  Endpoint | 28.8 (15.1) | 29.0 (13.7)

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | L-tetrahydropalmatine | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/32
Other Adverse Events (participants affected / at risk) | 29/29 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-tetrahydropalmatine (N=29) | Sugar Pill (N=32)
Severe Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | L-tetrahydropalmatine (N=29) | Sugar Pill (N=32)
Sedation (General disorders) | 9 | 10
Headache (General disorders) | 9 | 8
Nausea (Gastrointestinal disorders) | 7 | 9
Diarrhea (Gastrointestinal disorders) | 6 | 4
Dizziness (General disorders) | 9 | 3
Insomnia (General disorders) | 6 | 8
Vomiting (Gastrointestinal disorders) | 3 | 5
Abdominal Pain (General disorders) | 3 | 5
Constipation (General disorders) | 3 | 5
Malaise (General disorders) | 4 | 8
Restlessness (General disorders) | 2 | 7
Salivation (General disorders) | 5 | 9
Tinnitus (General disorders) | 1 | 7
Dry Mouth (General disorders) | 4 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02118610/Prot_SAP_000.pdf